CLINICAL TRIAL: NCT07216833
Title: Biomarker Driven Phase 1/1b Trial of Decitabine and Nivolumab in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Decitabine and Nivolumab in Participants With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyunghee Burkitt, DO, PhD (Other)
Responsible Party: Sponsor-Investigator, Kyunghee Burkitt, DO, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7324
Record Dates: First submitted 2025-10-08; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Head and Neck Squamous Cell Carcinoma
Keywords: Decitabine and Nivolumab
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Decitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Decitabine + Nivolumab (Experimental): Participants will receive 28-day cycles of decitabine followed by nivolumab for up to 35 cycles (up to 2 years) or until disease progression or other adverse event(s).
  Interventions: Drug: Decitabine; Drug: Nivolumab

INTERVENTIONS:
Drug: Decitabine — Participants will receive dose level 1 (DL1). If 2 of 3 participants experience dose limiting toxicity (DLT) on DL1, then the dose will be de-escalated to DL1-1. If 2 of 3 participants experience DLT on DL1-1, then no further de-escalation will occur and no additional participants will be enrolled.
  DL1: Intravenous (IV) administration of decitabine 20 mg/m2 from Days 1-5
  DL1-1: Intravenous (IV) administration of decitabine 20 mg/m2 from Days 1-4
Drug: Nivolumab — Nivolumab will be used as a fixed dose in combination with de-escalating dose levels (DL1, DL1-1) of decitabine.
  Participants will receive 480 mg of nivolumab on Day 8 every 4-week cycle.

SUMMARY:
This research study is for people who have recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) that has been confirmed by tissue or cell analysis and is considered incurable with local treatments. People who are eligible to receive anti-PD-L1 therapy as a first line treatment and whose primary tumor is located in the oral cavity, oropharynx, hypopharynx, or larynx, may be eligible to participate.

The purpose of this study is to evaluate the immunogenicity of decitabine in combination with nivolumab, and to evaluate the safety and tolerability of decitabine in combination with nivolumab and to determine the maximum tolerated dose.

Decitabine is a drug that is currently approved by the Food and Drug Administration (FDA) for the treatment of myelodysplastic syndrome (MDS). Decitabine is considered an investigational (experimental) drug in this study because it is not approved by the FDA for the treatment of HNSCC. Decitabine is a chemotherapy drug that works by targeting DNA methylation, a process that can restore normal function to genes that are involved in cell growth and differentiation. This can help reduce the growth of cancer cells.

Nivolumab is a drug that is approved by the FDA for the treatment of HNSCC, as well as other types of cancer. Nivolumab is an immunotherapy drug that works by helping the body's immune system recognize and attack cancer cells.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is the 6th most common cancer worldwide with approximately 60,000 people diagnosed each year in the United States. People with human papilloma virus (HPV)-positive HNSCC usually have a good prognosis, but HPV-negative people have about a 50% chance that their cancer will come back even after being treated. People who have recurrent or metastatic (R/M) HNSCC who are treated for their cancer tend to have an even worse prognosis, with a median overall survival of about 10 months. An anti-programmed-death-1 (anti-PD1) inhibitor called pembrolizumab was recently approved to treat people with R/M HNSCC. Another type of anti-PD1 inhibitor is a drug called nivolumab, which is also approved to treat people with R/M HNSCC. However, response rates to both pembrolizumab and nivolumab monotherapy are as low as 19% and 13.3% respectively. This shows that there are immune-evasive mechanisms present, meaning that tumor cells can more easily evade being detected and destroyed. Decitabine is a drug that may help anti-PD1 inhibitors like nivolumab better detect and destroy tumor cells. Previous research has shown that using a DNA methyltransferase inhibitor before giving a PD1 inhibitor to treat cancer can help the body's immune system more effectively kill cancer cells. Decitabine is a drug that is a type of DNA methyltransferase inhibitor. The purpose of this study is to evaluate the safety and tolerability of using decitabine in combination with nivolumab to treat HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed recurrent or metastatic HNSCC considered incurable by local therapies and eligible to receive anti-PD-L1 as first-line treatment (PD-L1 positive with combined positive score (CPS) 1 as evaluated in pre-screening).
* Participants must have primary tumor locations in following; oral cavity, oropharynx, hypopharynx, or larynx (nasopharynx is not allowed).
* No systemic therapy administered in the recurrent or metastatic setting (except for systemic therapy completed within 6 months or > 6 months if given as part of multimodal treatment for locally advanced disease).
* Participants must not have received prior treatment with immune checkpoint inhibitors.
* For primary site locally recurrent HNSCC, participants can provide archival tumor tissue not older than 3 months from a core or excisional biopsy for PD-L1 pre-screening using the PD-L1 IHC 22C3 pharmDx assay.
* For metastatic cancer patients, archival tumor tissue of distant metastatic lesion should not be older than 3 months from a core biopsy for PD-L1 pre-screening using the PD-L1 IHC 22C3 pharmDx assay.
* For primary site locally recurrent HNSCC, participants must have lesions amenable to obtain pre-treatment tumor biopsies in screening period after eligibility confirmation and before start of treatment and on-treatment tumor biopsies on C1D8 & C3D21 after start of treatment if lesions are still present at that time. If a recent archival biopsy is obtained within 3 months prior to start of treatment, this biopsy can be used as a pre-treatment biopsy.
* Participants should be ≥ 18 years of age
* Participants should have ECOG Performance status ≤ 2
* Participants must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dl
  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits (Gilbert's syndrome related elevated bilirubin is accepted as long as levels have been stable within last 3 months).
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Serum creatinine within normal institutional limits
* Women of child-bearing potential and sexually active men with female partners of child-bearing potential must agree to use a highly effective method of contraception beginning with the first dose of study therapy and for the duration of their participation in the study. This is expected for the entire duration of the study period through 6 months after the last dose. Highly effective methods of contraception include female sterilization (tubal ligation, bilateral oophorectomy, and/or hysterectomy); male sterilization (at least 6 months prior to screening); intrauterine device; and oral, injected, or implanted hormonal contraception AND barrier methods of contraception. Women of child-bearing potential must have documented negative pregnancy test prior to start of investigational treatment regimen. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with progressive disease within six months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Participants with history of severe immune related adverse effects from prior immunotherapy, except hypothyroidism clinically stable on hormone replacement treatment and controlled type 1 diabetes. All other endocrinopathies are excluded even if controlled with medications.
* Participants with Grade ≥ 3 infections within 4 weeks before the first study drug administration. Clinically active infections > Grade 1 within 2 weeks before the first study drug administration.
* Participants with previous or active myocarditis/myositis in history (independent of cause).
* Participants with pneumonitis, idiopathic pulmonary fibrosis, organizing, interstitial lung disease active or history of autoimmune disease. Autoimmune thyroid disease as well as other non-life-threatening autoimmune diseases such as vitiligo or autoimmune alopecia that don't require systemic immunosuppression are not excluded.
* Participants with known human immunodeficiency virus (HIV) infection, uncontrolled active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Participants with treatment with systemic immunosuppressant medications within 2 weeks before the first study drug administration. However, low-dose steroid use (prednisone equivalent <=10 mg daily) for other reasons is allowed.
* Participants receiving any other investigational agents.
* Participants with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with confirmed COVID-19. Participants with confirmed COVID-19 within 7 days prior to starting treatment will be excluded, however upon recovery with confirmation of negative COVID test, participant can be reconsidered for the study.
* Participants with a history of hypersensitivity to active or inactive excipients of decitabine or nivolumab or drugs with a similar chemical structure or class to either agent.

Participants with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics data on the effects of decitabine, as measured by change in global DNA methylation status | Day 1, Day 8
  DNA methylation will be measured pre- and post-decitabine administration and will be compared using Wilcoxon signed-rank test. Methylation analysis requires 500ng of isolated DNA and will be performed on the Illumina Infinium EPIC array.
Immunogenicity of decitabine in combination with nivolumab, as measured by change in immunologic biomarkers | Day 1, Day 8
  Changes in immunologic biomarkers will be correlated with changes in DNA methylation, measured pre- and post-decitabine administration. Immunologic biomarkers include PD-L1 expression (IHC), HLA Class I protein expression (IHC), TIL (tumor infiltrating lymphocytes, IHC and multiplex IF).
Safety and tolerability of decitabine in combination with nivolumab, as measured by number of adverse events | Up to 35 days post-treatment discontinuation (treatment may last up to 2 years)
  Participants will be evaluated for safety with a follow up visit approximately 28 (+/- 7) days after treatment discontinuation. The National Cancer Institute Common Terminology Criteria for Advanced events (NCI CTCAE) version 5 will be used for adverse event grading. Safety evaluation will be measured by reviewing the adverse event (AE) profile, clinical laboratory safety tests, vital signs, and ECG monitoring.
Maximum tolerated dose (MTD) | Through treatment period, up to 35 cycles (each cycle is 28 days) or up to 2 years
  MTD is defined as the dose level at which safety can be confirmed. If 2 or more out of 3 participants experienced a dose limiting toxicity (DLT), the dose will be de-escalated and evaluated for safety. MTD will be evaluated through the treatment period. Participants will receive treatment of up to 35 treatment cycles until disease progression or other adverse event(s).

SECONDARY OUTCOMES:
Objective response rate (ORR) | End (week 4) of every 3 cycles, up to 35 total cycles (each cycle is 28 days) or up to 2 years
  ORR is the percentage of participants whose cancer got better after treatment (i.e. the percentage of participants who had CR or PR, as defined below), and this will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
  Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of one or more new lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Overall survival (OS) | Until death, up to 2 years
  Overall survival (OS) is defined as the duration of time from start of treatment to time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghee Burkitt, DO, PhD, MS, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underline results in publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data included in the peer reviewed publication will be publicly available indefinitely. No raw data will be shared.
Access Criteria: A peer-reviewed publication will be made available according to the publishing journal's specifications. CCF personnel will not share study data apart from that which has been published publicly.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Ghoneim HE, Fan Y, Moustaki A, Abdelsamed HA, Dash P, Dogra P, Carter R, Awad W, Neale G, Thomas PG, Youngblood B. De Novo Epigenetic Programs Inhibit PD-1 Blockade-Mediated T Cell Rejuvenation. Cell. 2017 Jun 29;170(1):142-157.e19. doi: 10.1016/j.cell.2017.06.007. Epub 2017 Jun 22. PMID 28648661
- [Background] Pauken KE, Sammons MA, Odorizzi PM, Manne S, Godec J, Khan O, Drake AM, Chen Z, Sen DR, Kurachi M, Barnitz RA, Bartman C, Bengsch B, Huang AC, Schenkel JM, Vahedi G, Haining WN, Berger SL, Wherry EJ. Epigenetic stability of exhausted T cells limits durability of reinvigoration by PD-1 blockade. Science. 2016 Dec 2;354(6316):1160-1165. doi: 10.1126/science.aaf2807. Epub 2016 Oct 27. PMID 27789795